CLINICAL TRIAL: NCT01309399
Title: Early Effects of PTH on the Proximal Femur
Brief Title: Early Effects of Parathyroid Hormone (PTH) on the Proximal Femur
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Health Research, Inc. (Other)
Collaborators: Hospital for Special Surgery, New York (Other); National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Principal Investigator, Felicia Cosman, M.D., Medical Director, Clinical Research Center, Helen Hayes Hospital, Health Research, Inc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: 09-09; R01AR059204-01 (NIH)
Record Dates: First submitted 2011-03-04; First posted 2011-03-07 (Estimated); Last update posted 2016-11-23 (Estimated); Status verified 2016-11

CONDITIONS: Osteoporosis
Keywords: bone formation rate; total hip arthroplasty
MeSH Terms: conditions — Osteoporosis | interventions — Teriparatide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- teriparatide (Active Comparator): six weeks of teriparatide
  Interventions: Drug: Teriparatide
- placebo (Placebo Comparator): placebo identical in appearance to teriparatide
  Interventions: Other: placebo

INTERVENTIONS:
Drug: Teriparatide — six weeks of teriparatide
  Other Names: forteo
  Arms: teriparatide
Other: placebo — placebo
  Arms: placebo

SUMMARY:
Teriparatide is a potent osteoporosis medication that helps prevent fractures, however, the investigators know little about its effect on the hip. The investigators will evaluate hip bone samples from patients treated with teriparatide before undergoing hip replacement. The information will help us understand how teriparatide might help reduce hip fracture risk.

DETAILED DESCRIPTION:
Osteoporosis with consequent hip fractures causes substantial disability, morbidity and mortality. Teriparatide (TPTD), the aminoterminal fragment of parathyroid hormone (PTH), increases bone mineral density (BMD) and bone strength and reduces fracture incidence throughout the skeleton, but data confirming specific efficacy against hip fracture will never be available. Histomorphometric studies after 18-36 months of TPTD treatment show improvements in bone volume and structure in the iliac crest. Both biochemical and histomorphometric investigations of the iliac crest at very early time points (within 4-6 weeks of administration) show that bone formation is dramatically stimulated. Apart from the beneficial effect of TPTD on bone density and bone strength by finite element analysis at the hip, nothing is known about the mechanism of the effect of TPTD on the proximal femur. While BMD changes are smaller and slower in the hip in response to TPTD than in the spine, it is possible that stimulation of bone formation on the periosteal bone surface could result in expansion of bone size, obscuring the increase in non-invasively measured BMD. The current study will provide evidence for or against this possible TPTD-induced periosteal expansion. From a clinical perspective, it is unclear whether TPTD would be preferable to other osteoporosis medications, such as zoledronic acid, in patients at high risk for hip fracture. TPTD induced bone formation in the femur would be expected to improve bone strength and would provide a mechanistic basis for the use of TPTD in patients at high risk of hip fracture. The proposed project is the only practical and ethical way to obtain information on the effects of TPTD on bone formation in the proximal femur in humans. In patients undergoing total hip arthroplasty (THA) for degenerative joint disease, the hip samples of greatest interest are extracted routinely during the procedure. At the same time, an iliac crest biopsy can be taken with minimal added time and risk. The protocol has the following Specific Aims:

In patients undergoing elective, noncemented total hip arthroplasty (THA): 1. To determine the early effects of 1-34hPTH (teriparatide; TPTD 20 mcg) vs placebo, administered subcutaneously daily for 6 weeks, on histomorphometric indices of bone formation in cancellous and cortical bone of the proximal femur (femoral neck and intertrochanteric bone) and iliac crest. 2. To evaluate the association between changes in biochemical indices of bone turnover and histomorphometric indices of bone formation in the proximal femur (femoral neck and intertrochanteric bone) and iliac crest over 6 weeks of treatment with TPTD vs. placebo. 3. To determine if circulating osteoblast precursor cells increase over 6 weeks of treatment with TPTD vs Placebo and to compare the change in size of this osteoblast precursor pool with the change in a biochemical marker of bone formation and indices of bone formation in the femur and iliac crest.

ELIGIBILITY:
Inclusion Criteria:

* Age 50-90 years old.
* Male or postmenopausal (women who have had no menses for one year)
* Degenerative joint disease of the hip (osteoarthritis) requiring total hip arthroplasty, based on radiologic and clinical impression.

Exclusion Criteria:

* Any contraindications to use of TPTD.
* Age younger than 50, greater than 90 years old.
* Metabolic bone disease other than osteoporosis.
* History of hyperparathyroidism without surgical correction.
* Unexplained hypercalcemia.
* Paget's disease (or unexplained elevated bone alkaline phosphatase level).
* History of any metastatic cancer or osteosarcoma.
* Prior radiation treatment.
* Secondary hyperparathyroidism due to vitamin D deficiency or renal disease. Active hyperthyroidism or excessive thyroid hormone replacement (with TSH below normal range).

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-08; Primary Completion 2014-11 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Bone formation rate | 6 weeks
  At the time of surgery, the femoral neck and a small piece of bone will be obtained and measured for indices of bone formation in the femur and iliac crest in both placebo or teriparatide groups.

SECONDARY OUTCOMES:
Blood samples will be analyzed for indices of bone formation (serum P1NP) and resorption (serum CTX) after treatment with placebo or teriparatide Biochemical markers of bone | six weeks
  Blood samples will be analyzed for indices of bone formation (serum P1NP) and resorption (serum CTX) after treatment with placebo or teriparatide

CONTACTS AND LOCATIONS:
Overall Officials: Felicia Cosman, M.D., Principal Investigator — Helen Hayes Hospital
Locations (1):
- Helen Hayes Hospital, West Haverstraw, New York, United States